CLINICAL TRIAL: NCT06113003
Title: The Gut, Liver And Metabolome in Human Immunodeficiency Virus and Non Alcoholic Fatty Liver Disease
Acronym: GLAM HIV NAFLD
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Curtis Gabriel, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 231185
Record Dates: First submitted 2023-10-24; First posted 2023-11-02 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: HIV; Non-Alcoholic Fatty Liver Disease; Metabolic-Associated Steatotic Liver Disease
Keywords: HIV; NAFLD; MASLD; Fiber; Microbiome; Probiotic; Prebiotic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Prebiotics; Probiotics

STUDY DESIGN:
Intervention Model Description: Pre/Post Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Probiotic and Prebiotic Fiber (Experimental)
  Interventions: Dietary Supplement: Prebiotic; Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Prebiotic — Wheat dextrin fiber
Dietary Supplement: Probiotic — Probiotic packet

SUMMARY:
Persons with human immunodeficiency virus (HIV) have higher risk of developing fatty liver disease (NAFLD) than HIV-negative persons but the reasons for this discrepancy are not known. Changes in the intestinal microbiome may contribute to the development of NAFLD in persons with HIV (PWH) through impairment of barrier function of the intestinal wall and by producing metabolites that are harmful to the liver. This project will test the hypothesis that HIV-related NAFLD is associated with differences in the intestinal microbiome and that supplementation with probiotic and prebiotic fiber will lead to improvements in markers of NAFLD in PWH.

DETAILED DESCRIPTION:
Over 1.1 million people in the United States are living with human immunodeficiency virus (HIV). Liver disease is a leading cause of mortality in persons with HIV (PWH), and PWH suffer a disproportionate burden of non-alcoholic fatty liver disease (NAFLD). While the mechanisms underlying this disparity are not well understood, harmful changes in the intestinal microbiome ("dysbiosis") and increased bacterial product movement across the intestinal lining ("leaky gut") are implicated in the pathogenesis of NAFLD in HIV-negative persons. HIV infection has been shown to alter the intestinal microbiome and promote leaky gut; however, there are few data on the microbiome among PWH with NAFLD. Our overarching hypothesis is that intestinal dysbiosis in PWH promotes NAFLD through: 1) impairment of the barrier function of the intestinal lining causing translocation of proinflammatory bacterial products to the bloodstream and 2) alteration of plasma metabolites that promote NAFLD. Specifically, HIV-associated gut dysbiosis leads to reduction in the production of short chain fatty acids, which are essential for the maintenance of a healthy intestinal lining. A reduction in butyrate production leads to breakdown of the intestinal barrier, allowing for translocation of inflammatory bacterial products into the splanchnic vasculature and the liver. These products lead to inflammation and disruption of lipid metabolism in the liver causing lipid deposition in the liver. Additionally, dysbiosis in PWH leads to lower bacterial production of lipids necessary for fat metabolism in the liver leading to NAFLD. We will test these hypotheses in a single arm pre/post feasibility and efficacy trial of an intervention designed to restore a healthy gut microbiome in PWH with NAFLD (n=63). The study will assess the effects of a probiotic containing multiple strains of bacteria supporting butyrate synthesis and prebiotic fiber among PWH at risk of NAFLD (diagnosis of metabolic syndrome, elevated BMI or elevated transaminases) without history of current excessive alcohol use, viral hepatitis or other known liver diseases.

ELIGIBILITY:
Inclusion Criteria:

* One of the following:

  1. One or more of the components of metabolic syndrome, defined as:

     1. Diagnosis of diabetes: on medication for diabetes for at least 6 months, HbA1c >6.5%, or fasting glucose >99 mg/dL
     2. Elevated fasting triglycerides: >149 mg/dL or on medication for dyslipidemia
     3. Reduced HDL-C: <40 mg/dL in males, <50 mg/dL in females or on medication for dyslipidemia
     4. Elevated blood pressure: >129 mm Hg systolic and/or >84 mm Hg diastolic or on medication for hypertension
     5. Prior diagnosis of hepatic steatosis or NAFLD: hepatic steatosis noted on interpretation of clinical imaging, CT scan liver density of less than 58 HU, Fibroscan CAP score >238 dB/m, MRI-PDFF ≥5%, liver biopsy showing ≥5% triglyceride content
  2. Persistently abnormal transaminases: elevated liver enzymes defined by transaminases ≥1.5 upper limit of normal ([ULN] = 35 IU/mL) and/or gammaglutamyltransferase level ≥2 ULN (ULN = 60 IU/L) on 2 blood samples within at least a 3-month interval
  3. BMI ≥ 30 kg/m2
* Documented HIV infection
* On antiretroviral therapy for at least 18 months
* HIV-1 RNA <50 copies/ml for the prior 12 months
* CD4 count >350 cells/microliter for the prior 12 months
* Ability to be contacted by phone (home or cell)
* Access to a private (i.e. accessible only to participant and immediate family or roommates) refrigerator for 6 months
* Able and willing to comply with all study protocols and procedures

Exclusion Criteria:

* Not fluent in English
* Known allergy to the study product or its formulation
* Pregnant or planning to become pregnant within the next six months
* History of chronic diarrhea in the past three months
* Breastfeeding
* History of celiac disease
* Prior diagnosis of non-NAFLD liver disease including, but not limited to, Wilson Disease, hemochromatosis, autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, and alpha 1 antitrypsin deficiency
* On medications associated with secondary NAFLD including systemic corticosteroids, tamoxifen, methotrexate, nifedipine, history of cancer chemotherapy,
* Positive hepatitis C quant or on treatment for hepatitis C within the last 12 months
* History of cirrhosis or liver transplant
* AUDIT-C score ≥3 women and ≥4 in men
* History of inflammatory bowel disease
* History of all other GI surgery within the past 12 months
* Use of antibiotics in the past 30 days
* Metal shrapnel, MRI incompatible hardware or claustrophobia that would preclude MRI imaging
* Inability to participate in the study in the opinion of the participant's HIV treatment provider
* Use of prebiotic(s) including fiber supplements and/or probiotic(s) within the past 90 days
* Participant has history of hemicolectomy, colectomy, small bowel resection, bariatric surgery, gastric bypass surgery, or short bowel syndrome

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Plasma phosphatidylcholine | 24 weeks
  Plasma phosphatidylcholine abundance is measured

SECONDARY OUTCOMES:
Proton Density Fat Fraction | 24 weeks
  Hepatic steatosis is measured using magnetic resonance imaging proton density fat fraction
Simpson Index | 24 weeks
  The Simpson Index is a measure of intestinal bacterial diversity.
Soluble CD14 | 24 weeks
  Soluble CD14 is an indirect plasma markers of intestinal barrier function
Fatty Acid Binding Protein | 24 weeks
  Fatty acid binding protein is an indirect plasma markers of intestinal barrier function
CD163 | 24 weeks
  CD163 is an indirect plasma markers of intestinal barrier function
Firmicutes-to-Bacteroidetes Ratio | 24 weeks
  The Firmicutes-to-Bacteroidetes ratio is a measure of intestinal bacterial diversity.
Shannon Index | 24 weeks
  The Shannon Index is a measure of intestinal bacterial diversity.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD outside of VUMC study team.